CLINICAL TRIAL: NCT01452243
Title: Prevention of Falls and Fractures in Old People by Administration of Calcium and Vitamin D. Randomized Clinical Trial (ANVITAD)
Brief Title: Prevention of Falls and Fractures in Old People by Administration of Calcium and Vitamin D. Randomized Clinical Trial
Acronym: ANVITAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gerencia de Atención Primaria, Albacete (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006001
Record Dates: First submitted 2011-10-09; First posted 2011-10-14 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Fall; Fractures
Keywords: Vitamin D; Calcium; Elderly
MeSH Terms: conditions — Fractures, Bone | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcium and vitamin D (Experimental): The pharmacological intervention will be the daily administration of chewable tablets containing vitamin D and calcium.
  Interventions: Drug: Vitamin D and calcium suplementation

INTERVENTIONS:
Drug: Vitamin D and calcium suplementation — The pharmacological intervention will be the daily administration of chewable tablets containing 800 IU of vitamin D and 1200 mg of calcium. They will be administered over 2 years during the months of November to April in order to avoid the influence of sunlight.

SUMMARY:
The first objective is to determine the efficacy of calcium and vitamin D supplementation at doses of 1200 mg and 800 IU, respectively, to reduce the incidence of falls and fractures in non-institutionalized elderly people.

The second objective is to measure and compare treatment groups (calcium and vitamin D vs placebo) as regards muscle strength and musculoskeletal function, bone mineral density, calcidiol level and treatment safety.

DETAILED DESCRIPTION:
Background:

There are many studies that associate vitamin D serum levels in older persons with muscle strength, physical performance and risk of fractures and falls. However, current evidence is insufficient to make a general recommendation for administrating calcium and vitamin D to older persons. The objective of this study is to determine the effectiveness of calcium and vitamin D supplementation in improving musculoskeletal function and decreasing the number of falls in person aged over 65 years.

Design:

Phase III, randomized, double blind, placebo-controlled trial to evaluate the efficacy of already marketed drugs in a new indication. It will be performed at Primary Care doctor visits at several Healthcare Centers in different Spanish Health Areas. A total of 704 non-institutionalized subjects aged 65 years or older will be studied (sample size calculated for a statistical power of 80%, alpha error 0.05, annual incidence of falls 30% and expected reduction of 30% to 20% and expected loss to follow up of 20%). The test drug containing 800 IU of vitamin D and 1000 mg of calcium will be administered daily. The control group will receive a placebo. The subjects will be followed up over two years. The primary variable will be the incidence of spontaneous falls. The secondary variables will include: consequences of the falls (fractures, need for hospitalization), change in calcidiol plasma levels and other analytical determinations (transaminases, PTH, calcium/phosphorous, albumin, creatinine, etc.), change in bone mass by densitometry, change in muscle strength in the dominant hand and change in musculoskeletal strength, risk factors for falls, treatment compliance, adverse effects and socio-demographic data.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 65 years with normal renal function
* Normal transaminase levels
* Normal calcium blood levels
* Not homebound (not immobilized) nor in socio-healthcare institutions.

Exclusion Criteria:

* Need for medical treatment with calcium or vitamin D
* Hypersensitivity to or contraindication for calcium or vitamin D
* Medical treatment that includes calcium or vitamin D
* Physical disability that impedes their collaboration
* Taking thiazide diuretics
* Oral anticoagulants
* Hormone replacement therapy
* Digitalis drugs
* Anticonvulsants or barbiturates
* Having any of the following diseases:

  * Lithiasis
  * Renal impairment (serum creatinine >1.4 mg/dl)
  * Hypo or hyperthyroidism
  * Paget's disease
  * Chronic liver disease
  * Tumors
  * Sarcoidosis
  * Impaired intestinal absorption or chronic alcoholism (>40 g/day).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 704 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of spontaneous falls. | 24 months.
  The primary variable will be the incidence of spontaneous falls according to the FICSIT (Frailty and Injury: Cooperative Study of Intervention Techniques) definition: "Unintentionally coming to rest on the ground, floor, or other lower level. Coming to rest against furniture or a wall was not counted as a fall".

SECONDARY OUTCOMES:
Consequence of falls. | 24 months.
  Bone fractures at any location, need for healthcare, need for hospitalization, bed-ridden.
Change in calcidiol [25(OH)D3] plasma levels | 18 months.
  Determined by RIA (Vitamin D deficiency is defined as a calcidiol plasma level lower than 10ng/ml).
Change in bone mass (bone density or mineral content). | 24 months.
  By densitometry (risk of fracture). Osteoporosis will be diagnosed based on a densitometry T-score of less than 2.5 in the vertebral column, according to WHO criteria.
Change in muscle strength in the dominant hand. | 24 months
  Determined by dyanometry (with a mean of 3 attempts to obtain a muscle strength measurement).
Changes in musculoskeletal function. | 24 months
  By the timed up and go test (the elderly person gets up from a chair with arms, walks three meters, turns round, walks back and sits down again). Taking more than 20 seconds indicates a high risk for falls.
Serious adverse events or any other adverse event. | 24 months.
  An adverse event is considered as any untoward medical occurrence in any patient included in the study which does not necessarily have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús López-Torres, Hidalgo, Principal Investigator — Research Unit. Primary Care Head Office of Albacete; Ignacio Párraga Martínez, Dr., Study Chair — Research Unit. Primary Care Head Office of Albacete; Beatriz Navarro Bravo, Dr., Study Chair — Research Unit. Primary Care Head Office of Albacete; Fernando Andrés Pretel, Dr., Study Chair — Research Unit. Primary Care Head Office of Albacete
Locations (1):
- Research Unit. Primary Care Head Office of Albacete, Albacete, Albacete, Spain

REFERENCES:
- [Background] Bischoff HA, Stahelin HB, Dick W, Akos R, Knecht M, Salis C, Nebiker M, Theiler R, Pfeifer M, Begerow B, Lew RA, Conzelmann M. Effects of vitamin D and calcium supplementation on falls: a randomized controlled trial. J Bone Miner Res. 2003 Feb;18(2):343-51. doi: 10.1359/jbmr.2003.18.2.343. PMID 12568412
- [Background] Bischoff-Ferrari HA, Willett WC, Wong JB, Giovannucci E, Dietrich T, Dawson-Hughes B. Fracture prevention with vitamin D supplementation: a meta-analysis of randomized controlled trials. JAMA. 2005 May 11;293(18):2257-64. doi: 10.1001/jama.293.18.2257. PMID 15886381
- [Background] Campbell AJ, Robertson MC, Gardner MM, Norton RN, Tilyard MW, Buchner DM. Randomised controlled trial of a general practice programme of home based exercise to prevent falls in elderly women. BMJ. 1997 Oct 25;315(7115):1065-9. doi: 10.1136/bmj.315.7115.1065. PMID 9366737
- [Background] Chapuy MC, Arlot ME, Duboeuf F, Brun J, Crouzet B, Arnaud S, Delmas PD, Meunier PJ. Vitamin D3 and calcium to prevent hip fractures in elderly women. N Engl J Med. 1992 Dec 3;327(23):1637-42. doi: 10.1056/NEJM199212033272305. PMID 1331788
- [Background] Chapuy MC, Pamphile R, Paris E, Kempf C, Schlichting M, Arnaud S, Garnero P, Meunier PJ. Combined calcium and vitamin D3 supplementation in elderly women: confirmation of reversal of secondary hyperparathyroidism and hip fracture risk: the Decalyos II study. Osteoporos Int. 2002 Mar;13(3):257-64. doi: 10.1007/s001980200023. PMID 11991447
- [Background] del Campo MT, Aguado P, Martinez ME. [Vitamin D and bone health: is there a need to review supplementation in osteoporosis risk population?]. Med Clin (Barc). 2005 Dec 3;125(20):788-93. doi: 10.1016/s0025-7753(05)72191-6. Spanish. PMID 16373031
- [Background] Dhesi JK, Bearne LM, Moniz C, Hurley MV, Jackson SH, Swift CG, Allain TJ. Neuromuscular and psychomotor function in elderly subjects who fall and the relationship with vitamin D status. J Bone Miner Res. 2002 May;17(5):891-7. doi: 10.1359/jbmr.2002.17.5.891. PMID 12009020
- [Background] Gillespie WJ, Avenell A, Henry DA, O'Connell DL, Robertson J. Vitamin D and vitamin D analogues for preventing fractures associated with involutional and post-menopausal osteoporosis. Cochrane Database Syst Rev. 2001;(1):CD000227. doi: 10.1002/14651858.CD000227. PMID 11279685
- [Background] Janssen HC, Samson MM, Verhaar HJ. Vitamin D deficiency, muscle function, and falls in elderly people. Am J Clin Nutr. 2002 Apr;75(4):611-5. doi: 10.1093/ajcn/75.4.611. PMID 11916748
- [Background] Latham NK, Anderson CS, Reid IR. Effects of vitamin D supplementation on strength, physical performance, and falls in older persons: a systematic review. J Am Geriatr Soc. 2003 Sep;51(9):1219-26. doi: 10.1046/j.1532-5415.2003.51405.x. PMID 12919233
- [Background] Lips P, Graafmans WC, Ooms ME, Bezemer PD, Bouter LM. Vitamin D supplementation and fracture incidence in elderly persons. A randomized, placebo-controlled clinical trial. Ann Intern Med. 1996 Feb 15;124(4):400-6. doi: 10.7326/0003-4819-124-4-199602150-00003. PMID 8554248
- [Background] NIH Consensus Development Panel on Osteoporosis Prevention, Diagnosis, and Therapy. Osteoporosis prevention, diagnosis, and therapy. JAMA. 2001 Feb 14;285(6):785-95. doi: 10.1001/jama.285.6.785. PMID 11176917
- [Background] Pfeifer M, Begerow B, Minne HW. Vitamin D and muscle function. Osteoporos Int. 2002 Mar;13(3):187-94. doi: 10.1007/s001980200012. PMID 11991436
- [Background] Simon J, Leboff M, Wright J, Glowacki J. Fractures in the elderly and vitamin D. J Nutr Health Aging. 2002;6(6):406-12. PMID 12459891
- [Background] Vallecillo G, Diez A, Carbonell J, Gonzalez Macias J. [Treatment of osteoporosis with calcium and vitamin D. Systematic review]. Med Clin (Barc). 2000 Jun 10;115(2):46-51. doi: 10.1016/s0025-7753(00)71461-8. Spanish. PMID 10934692
- [Background] van der Wielen RP, Lowik MR, van den Berg H, de Groot LC, Haller J, Moreiras O, van Staveren WA. Serum vitamin D concentrations among elderly people in Europe. Lancet. 1995 Jul 22;346(8969):207-10. doi: 10.1016/s0140-6736(95)91266-5. PMID 7616799
- [Background] Zamboni M, Zoico E, Tosoni P, Zivelonghi A, Bortolani A, Maggi S, Di Francesco V, Bosello O. Relation between vitamin D, physical performance, and disability in elderly persons. J Gerontol A Biol Sci Med Sci. 2002 Jan;57(1):M7-11. doi: 10.1093/gerona/57.1.m7. PMID 11773206
- [Background] Zittermann A. Vitamin D in preventive medicine: are we ignoring the evidence? Br J Nutr. 2003 May;89(5):552-72. doi: 10.1079/BJN2003837. PMID 12720576
- [Derived] Lopez-Torres Hidalgo J; ANVITAD Group. Prevention of falls and fractures in old people by administration of calcium and vitamin D, randomized clinical trial. BMC Public Health. 2011 Dec 9;11:910. doi: 10.1186/1471-2458-11-910. PMID 22151975